CLINICAL TRIAL: NCT03231306
Title: A Phase II Study of Binimetinib in Children and Adults With NF1 Associated Plexiform Neurofibromas (PNOC010)
Brief Title: Phase II Study of Binimetinib in Children and Adults With NF1 Plexiform Neurofibromas
Acronym: NF108-BINI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Array BioPharma (Industry); Pacific Pediatric Neuro-Oncology Consortium (Other)
Responsible Party: Principal Investigator, Bruce Korf, MD, Principal Investigator, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-170616001; 516027 (Other Grant/Funding Number: Pfizer Inc., U.S. Pharmaceuticals Group)
Record Dates: First submitted 2017-07-21; First posted 2017-07-27 (Actual); Results first posted 2025-05-02 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Neurofibromatosis Type 1; Plexiform Neurofibroma
Keywords: Neurofibroma, Plexiform; Genes, Neurofibromatosis; Peripheral nerve tumors; Neurofibromatosis 1; Neurofibromas
MeSH Terms: conditions — Neurofibromatosis 1; Neurofibroma, Plexiform; Neurofibromatoses; Peripheral Nervous System Neoplasms; Neurofibroma | interventions — binimetinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Open label study of Binimetinib (MEK162) (Experimental): Subjects (≥ 18 years) (Stratum A) will receive a course of binimetinib by mouth twice a day (12 hours apart) of 45 mg/dose. Duration of each course is 4 weeks. After 8 courses, subjects will receive additional courses if MRI results showed at least 15% reduction in volume of the target tumor. Subjects can continue on therapy and will be evaluated at the end of 12 courses. Subjects who have ≥ 20% reduction in volume of the target tumor according to the MRI results can continue therapy up to an additional year (maximum of 24 total courses). Subjects who have not met the tumor reduction at the specified times will be removed from the study therapy. Subjects will be carefully monitored for toxicities associated with binimetinib.
  Recruitment of subjects 1 - 17 years of age (Stratum B) is currently available. The pediatric maximum tolerated dose (MTD) of binimetinib the pediatric patients (Statum B) was established by a phase 1 study (NCT022).
  Interventions: Drug: Binimetinib

INTERVENTIONS:
Drug: Binimetinib — Adult subjects (18 years and older) will receive binimetinib by mouth twice daily of 45mg/dose. Pediatric subjects (1-17 years of age) are being treated on the pediatric MTD established by a phase I study (NCT02285439).
  Other Names: MEK162 or ARRY-438162

SUMMARY:
This is a phase II open label study that will evaluate children ≥ 1 year of age and adults with neurofibromatosis type 1 (NF1) and plexiform neurofibromas treated with the MEK inhibitor, binimetinib. The primary objective is to determine if there is an adequate level of disease responsiveness to binimetinib in children and adults with NF1 and inoperable plexiform neurofibromas. The objective response to binimetinib is defined as ≥ 20% decrease in tumor volume reduction by 12 courses.

DETAILED DESCRIPTION:
Patients ≥ 1 year with progressive NF1 and PN(s) by serial imaging or causing significant morbidity and that can be analyzed by volumetric MRI are eligible for this study. Initially, the study will open to adult patients,18 years and older, (Stratum A). The pediatric patients (Statum B) will be receive the pediatric maximum tolerated dose (MTD) of binimetinib that is currently being established in an ongoing phase 1 study (NCT02285439). For adult subjects, binimetinib (established adult RP2D) is taken orally twice a day. Dosing will be continuous, with 28 days defined as a course and will continue for a total of 24 courses or until one of the Off Treatment or Off Study criteria are met. Subjects will undergo volumetric assays of their targeted PN using MRI after every 4 courses for the first year and then every 6 courses. MRI review of the volumetric assays will occur centrally under the guidance of Dr. Dombi at NCI. Subjects may receive additional courses beyond course 8 only if there is at least a 15% reduction in volume of the target tumor, as measured from baseline. Treatment beyond course 12 will be only be given to those subjects who achieve a response of ≥ 20% tumor shrinkage by volumetric analysis and can continue on therapy up to an additional year for a maximum of 24 total courses. For those who respond to binimetinib after 12 courses, an MRI scan of the target lesion must be performed at 4 and 12 months after stopping drug in order to determine whether response is maintained post-therapy. Subjects will be carefully monitored for development of binimetinib associated toxicities. Subjects will be removed from the study for significant toxicity, treatment delay of ≥ 21 days, or objective progression of tumor growth by ≥ 20% by volumetric analysis at any time.

The investigational nature and objectives of this trial, the procedures and treatment involved, the risks, discomforts, and benefits, and potential alternatives therapies will be carefully explained to the subject and/or subject's parent(s) or guardian by the site Principal Investigator or designated associate investigator. A signed informed consent document will be obtained prior to determining eligibility and entry criteria to this trial. Subjects entered on this trial will be treated with therapeutic intent and response to therapy will be closely monitored. This protocol involves greater than minimal risk but presents the potential for direct benefit to individual subjects.

Schedule of study evaluations are summarized below:

Pre-Study (Eligibility Screening):

* Physical assessment, vital signs and neurological exam
* Complete medical history including past and current medical conditions, treatments, and surgeries.
* Karnofsky/Lansky performance status to assess of your ability to perform everyday tasks
* Review of current medications
* Blood draw (about two tablespoons) for routine safety tests
* Serum or urine pregnancy test for females of childbearing age
* Eye exam
* Electrocardiogram (ECG) and echocardiogram (ECHO) or multigated acquisition (MUGA) scan of your heart
* MRI of neurofibroma tumors
* Functional evaluation: Depending on the location of your plexiform neurofibroma, specific functional assessments will be performed. The functional assessments may include a 6-Minute Walk-Test if you have a plexiform neurofibroma affecting your legs or airway, evaluation of muscle strength and range of motion if you have plexiform neurofibroma affecting your arms or legs, and/or grooved pegboard test if you have plexiform neurofibroma affecting your hands. The study team will review all evaluations that apply to you in detail
* Completion of health-related questionnaires on quality of life, pain assessment, bowel and bladder dysfunction, and PN symptom checklist (upon study entry)
* Photography of visible PN (optional)

End of course 1, 2, 3, 4, 6, 8, 10, 12, 15, 18, 21, and 24:

* Medical history update and hospitalization since last study visit
* Physical assessment, vital signs, and neurological exam
* Karnofsky/Lansky performance status to assess your ability to perform everyday tasks
* Review of your medication diary and any side effects you may be experiencing
* Review of current medications
* Blood draw (about two tablespoons) for routine safety tests
* Serum or urine pregnancy test for females of childbearing age

End of course 4, 8, 12, 18, and 24:

* Eye exam
* MRI of neurofibromas
* ECHO and ECG
* Functional evaluation: (see description above)
* Completion of health-related questionnaires on quality of life, pain assessment, bowel and bladder dysfunction, and PN symptom checklist
* Photography of visible PN (optional): If you agree to take part, photographs of visible PN will be taken. Photos will be taken before treatment and then after cycles 4, 8, 12, 18, and 24.

End of course 1 and 4:

• Blood draw (about one tablespoon) for cytokine studies (optional)

End of Treatment Visit (this is an additional visit if the visit is not within the specified times mentioned above):

* Physical assessment, vital signs and neurological exam
* Medical history update and hospitalization since last study visit
* Karnofsky/Lansky performance status to assess of your ability to perform everyday tasks
* Review of your medication diary and any side effects you may be experiencing
* Review of current medications
* Blood draw (about two tablespoons) for routine safety tests
* Serum or urine pregnancy test for females of childbearing age
* Eye exam
* Electrocardiogram (ECG) and ECHO or multigated acquisition (MUGA) scan of your heart
* MRI of neurofibroma tumors (for those who respond to binimetinib after 12 courses, an MRI at 4 and 12 months after stopping drug)
* Functional evaluation: (see description above)
* Completion of health-related questionnaires on quality of life, pain assessment, bowel and bladder dysfunction, and PN symptom checklist
* Photography of visible PN (optional)

The sample size is 20 subjects for each adult and children cohorts with a minimum target of 17 evaluable subjects per cohort. Evaluable is defined as: any subjects who received ≥ one dose of binimetinib and had a ≥ Grade 3 binimetinib associated toxicity, or in absence of a ≥ Grade 3 toxicity, any subjects who completed one full course of therapy; subjects who have completed at least two courses of therapy and had their first follow-up MRI evaluation except for discovery of a target tumor other than a PN; and any subjects who has at least two samples drawn for plasma cytokines/growth factors, one at baseline and at least one other after starting therapy.

Data Safety Monitoring Board (DSMB) and a Medical Monitor have been established for this study for the purpose of ensuring data compliance and regular monitoring. An early stopping rules have been defined within the protocol. The early stopping rule will invoked for both Strata separately to potentially prevent accrual subjects onto the study in the event that binimetinib is associated with a higher than acceptable rate of dose-limiting toxicity (DLT) requiring removal from study (10% or higher) during the first 2 courses. Toxicity will be continuously monitored. If at any time >2 of the first 10 subjects or 4 or more of the first 15 total subjects are removed for toxicity, then accrual will be stopped until the DSMB reviews the safety and efficacy data for the study. Based on the review, the DSMB can either recommend termination of the study or reopen recruitment. The Medical Monitor is a qualified physician who is not associated with this protocol and is a member of the DSMB. The Medical Monitor may perform oversight functions duties: may discuss the research protocol with the investigators, interview human subjects, and consult with others outside of the study about the research; shall have the authority to stop the research protocol in progress, remove individual subjects from protocol, and take whatever steps are necessary to protect the safety and well being of human subjects until the Institutional Review Board (IRB) can assess the monitor's report; and shall have the responsibility to promptly report the observation and findings to the IRB or other designated official/organization. The Medical Monitor is specifically required to review and provide written report of all unanticipated problems involving risk to subjects or others and serious adverse events.

In addition, as part of the Data Safety Monitoring Plan, the Study Chairs and the NF Consortium Clinical Research Nurse Manager will review subject eligibility, study progress, safety issues, protocol deviations and adverse events. Monthly reports will be generated by the NF Consortium Data Management Center to assess completeness of data. Monthly phone conferences will take place between NF Consortium Operations Center and the Protocol Team to address data issues.

The sample size for this trial is based on safety and feasibility factors. The data needed for safety is based on risk versus benefit, and for feasibility, we expect at least efficacy of 25% response rate. For safety reasons, subjects who do not achieve at least 15% reduction in volume of target tumor after 8 courses will be discontinued from the trial, as the likelihood of achieving a 20% reduction in tumor volume by 12 months is minimal. Safety analysis set will be described and summarized based on information regarding study treatment administrations, drug dosing and course compliance, and safety variables (e.g. adverse events/serious adverse events). All analyses for outcome results will be based on evaluable subjects. Given the difference in the clinical behavior of PN in the adults and pediatric subjects, the adult and children stratum will be analyzed independently.

ELIGIBILITY:
Inclusion Criteria

* Clinical diagnosis of NF1 using the NIH Consensus Conference criteria OR a documented constitutional NF1 mutation
* Plexiform neurofibroma(s) that are progressive or causing significant morbidity
* Presence of new plexiform neurofibroma on MRI or CT (documented by comparison with prior MRI or CT)
* Measurable plexiform neurofibroma(s) amenable to volumetric MRI analysis. Tumors must be at least 3 mL in volume (most PNs 3 cm in longest diameter will meet this criteria)
* Patients must be ≥ 18 years of age at the time of enrollment.
* Performance Level: Karnofsky or Lansky ≥ 50%. If unable to walk due to paralysis, but in a wheelchair, patients will be considered ambulatory for the purpose of assessing the performance level
* Ability to swallow capsules/tablets
* Ability to comply with follow up procedures
* The effects of binimetinib on the developing human fetus are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and 3 months after completion of binimetinib administration. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
* Negative urine or serum β-HCG test (females of childbearing potential only).

Prior Therapy:

* Patients are eligible if complete resection of a plexiform neurofibroma with acceptable morbidity is not feasible, or if a subject with surgical option refuses surgery,
* Patients who underwent surgery for a progressive plexiform neurofibroma will be eligible to enter the study after the surgery, provided the plexiform neurofibroma was incompletely resected and is evaluable by volumetric analysis.
* Patients previously treated for a plexiform neurofibroma or other tumor/malignancy, but must have fully recovered from the acute toxic effects of all prior chemotherapy or radiotherapy prior to entering this study.
* Must not have received myelosuppressive chemotherapy within 3 weeks of entry onto this study.
* At least 7 days since the completion of therapy with a hematopoietic growth factor that supports platelet, red or white cell number or function.
* At least 4 weeks since the completion of therapy with a biologic anti-neoplastic agent. For agents that have known adverse events occurring beyond 14 days after administration, this period must be extended beyond the time during which adverse events are known to occur.
* Patients must not have received an investigational drug within 4 weeks.
* Patients with endocrine deficiencies are allowed to receive physiologic or stress doses of steroids, if necessary.
* Radiation ≥ 6 months from involved field radiation to index plexiform neurofibroma(s), ≥ 6 weeks must have elapsed if patient has received radiation to areas outside index plexiform neurofibroma(s). Patients who have received radiation to the orbit at any time are excluded.
* At least 3 weeks since undergoing any major surgery and must be recovered from effects of surgery.

Organ Function Requirements:

* Adequate bone marrow function defined as:

  * Peripheral absolute neutrophil count (ANC) ≥ 1500/µL
  * Platelet count ≥ 100,000/µL (transfusion independent, defined as not receiving platelet transfusions for at least 7 days prior to enrollment)
  * Hemoglobin ≥ 10.0 gm/dL without transfusions.
* Adequate renal function defined as:

  * Maximum serum creatinine based on age/gender or a creatinine clearance or radioisotope GFR ≥ 70 ml/min/1.73 m²
* Adequate liver function defined as:

  * Bilirubin (sum of conjugated + unconjugated) ≤ 1.5 x upper limit of normal (ULN) for age
  * SGPT (ALT) ≤ 2.5 x upper limit of normal (ULN) for age
  * Serum albumin ≥ 2 g/dL
* Adequate cardiac function defined as:

  * Left ventricular fractions (LVEF) ≥ 50% as determined by a multigated acquisition (MUGA) scan or echocardiogram
  * QTc interval ≤ 480 ms.

Exclusion Criteria

* Chronic treatment with systemic steroids or another immunosuppressive agent.
* Evidence of an active optic glioma or other low-grade glioma, requiring treatment with chemotherapy or radiation therapy. Patients not requiring treatment are eligible for this protocol.
* Patients with malignant glioma, malignant peripheral nerve sheath tumor, or other malignancy requiring treatment in the last 12 months.
* Patients who have received radiation to the orbit at any time previously.
* Ophthalmologic conditions:

  * Current or past history of central serous retinopathy
  * Current or past history of retinal vein occlusion
  * Known intraocular pressure (IOP) > 21 mmHg (or ULN adjusted by age) or uncontrolled glaucoma (irrespective of IOP). Patients with known glaucoma and increased IOP who do not have meaningful vision (light perception only or no light perception) and are not experiencing pain related to the glaucoma, may be eligible after review. Patients with orbital plexiform neurofibromas should have IOP measured prior to enrollment.
  * Patients with any other significant abnormality on ophthalmic examination will be reviewed for potential eligibility.
  * Ophthalmological findings secondary to long-standing optic pathway glioma (such as visual loss, optic nerve pallor or strabismus) or long-standing orbito-temporal PN (such as visual loss, strabismus) will NOT be considered a significant abnormality for the purposes of the study
* Uncontrolled arterial hypertension despite medical treatment defined as CTCAE grade 3 or higher.
* Impaired cardiovascular function or clinically significant cardiovascular diseases, including:

  * History of acute coronary syndromes (including myocardial infarction, unstable angina, coronary artery bypass grafting, coronary angioplasty, or stenting) < 6 months prior to screening
  * Symptomatic chronic heart failure, history or current evidence of clinically significant cardiac arrhythmia and/or conduction abnormality < 6 months prior to screening except atrial fibrillation and paroxysmal supraventricular tachycardia
* Other concurrent severe and/or uncontrolled medical disease, which could compromise participation in the study (e.g. uncontrolled diabetes, uncontrolled hypertension, severe infection, severe malnutrition, chronic liver or renal disease, active upper GI tract ulceration, congestive heart failure, etc.)
* Subjects who have an uncontrolled infection.
* Known positive serology for HIV (human immunodeficiency virus), active hepatitis B, and/or active hepatitis C infection.
* Impairment of gastrointestinal function or gastrointestinal disease (e.g. ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome or small bowel resection).
* History of Gilbert's syndrome or patients who are known to be homozygous for UGT1A1 (7/7).
* Patients who have neuromuscular disorders that are associated with elevated CK (e.g., inflammatory myopathies, muscular dystrophy, amyotrophic lateral sclerosis, spinal muscular atrophy)
* Patients who are planning to embark on a new strenuous exercise regimen after first dose of study treatment. NB: muscular activities, such as strenuous exercise, that can result in significant increases in plasma CK levels should be avoided while on binimetinib treatment.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to binimetinib.
* Women who are pregnant or breastfeeding.
* Any other condition that would contraindicate, in the Investigator's judgement, the patient's participation in the clinical study due to safety concerns or compliance with clinical study procedures, e.g. infection/inflammation, intestinal obstruction, unable to swallow medication, social/ psychological issues, etc.
* History of noncompliance to medical regimens.
* Patients unwilling to or unable to comply with the protocol, or who in the opinion of the investigator may not be able to comply with the safety monitoring requirements of the study.
* Prior treatment with a MEK inhibitor of any kind.

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2017-11-28 (Actual); Primary Completion 2024-04-17 (Actual); Study Completion 2024-04-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Korf, MD, PhD, Study Chair — University of Alabama at Birmingham
Locations (22):
- United States (22):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Children's Hospital of Los Angeles, Los Angeles, California
  - University of California at Los Angeles, Los Angeles, California
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - University of California, San Diego - Rady Children's Hospital, San Diego, California
  - University of California, San Francisco, San Francisco, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Lurie Children's Hospital of Chicago, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - Johns Hopkins University, Baltimore, Maryland
  - National Institute of Health - National Cancer Institute, Bethesda, Maryland
  - Boston Children's Hospital / Dana Farber Cancer Institute / Massachusetts General Hospital, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - New York University Medical Center, New York, New York
  - Cinncinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Ohio State University, Columbus, Ohio
  - Oregon Health and Science University Hospital, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Utah, Salt Lake City, Utah
  - University of Washington - Seattle Children's Hospital, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wu J, Williams JP, Rizvi TA, Kordich JJ, Witte D, Meijer D, Stemmer-Rachamimov AO, Cancelas JA, Ratner N. Plexiform and dermal neurofibromas and pigmentation are caused by Nf1 loss in desert hedgehog-expressing cells. Cancer Cell. 2008 Feb;13(2):105-16. doi: 10.1016/j.ccr.2007.12.027. PMID 18242511
- [Background] Kebudi R, Cakir FB, Gorgun O. Interferon-alpha for unresectable progressive and symptomatic plexiform neurofibromas. J Pediatr Hematol Oncol. 2013 Apr;35(3):e115-7. doi: 10.1097/MPH.0b013e318270cd24. PMID 23042022
- [Background] Citak EC, Oguz A, Karadeniz C, Okur A, Memis L, Boyunaga O. Management of plexiform neurofibroma with interferon alpha. Pediatr Hematol Oncol. 2008 Sep;25(7):673-8. doi: 10.1080/08880010802315983. PMID 18850480
- [Background] Jakacki RI, Dombi E, Potter DM, Goldman S, Allen JC, Pollack IF, Widemann BC. Phase I trial of pegylated interferon-alpha-2b in young patients with plexiform neurofibromas. Neurology. 2011 Jan 18;76(3):265-72. doi: 10.1212/WNL.0b013e318207b031. PMID 21242495
- [Background] Widemann BC, Arceci RJ, Jayaprakash N, Fox E, Zannikos P, Goodspeed W, Goodwin A, Wright JJ, Blaney SM, Adamson PC, Balis FM. Phase 1 trial and pharmacokinetic study of the farnesyl transferase inhibitor tipifarnib in children and adolescents with refractory leukemias: a report from the Children's Oncology Group. Pediatr Blood Cancer. 2011 Feb;56(2):226-33. doi: 10.1002/pbc.22775. Epub 2010 Sep 21. PMID 20860038
- [Background] Widemann BC, Salzer WL, Arceci RJ, Blaney SM, Fox E, End D, Gillespie A, Whitcomb P, Palumbo JS, Pitney A, Jayaprakash N, Zannikos P, Balis FM. Phase I trial and pharmacokinetic study of the farnesyltransferase inhibitor tipifarnib in children with refractory solid tumors or neurofibromatosis type I and plexiform neurofibromas. J Clin Oncol. 2006 Jan 20;24(3):507-16. doi: 10.1200/JCO.2005.03.8638. PMID 16421428
- [Background] Babovic-Vuksanovic D, Widemann BC, Dombi E, Gillespie A, Wolters PL, Toledo-Tamula MA, O'Neill BP, Fox E, MacDonald T, Beck H, Packer RJ. Phase I trial of pirfenidone in children with neurofibromatosis 1 and plexiform neurofibromas. Pediatr Neurol. 2007 May;36(5):293-300. doi: 10.1016/j.pediatrneurol.2007.01.009. PMID 17509460
- [Background] Babovic-Vuksanovic D, Ballman K, Michels V, McGrann P, Lindor N, King B, Camp J, Micic V, Babovic N, Carrero X, Spinner R, O'Neill B. Phase II trial of pirfenidone in adults with neurofibromatosis type 1. Neurology. 2006 Nov 28;67(10):1860-2. doi: 10.1212/01.wnl.0000243231.12248.67. Epub 2006 Oct 11. PMID 17035676
- [Background] Kim A, Dombi E, Tepas K, Fox E, Martin S, Wolters P, Balis FM, Jayaprakash N, Turkbey B, Muradyan N, Choyke PL, Reddy A, Korf B, Widemann BC. Phase I trial and pharmacokinetic study of sorafenib in children with neurofibromatosis type I and plexiform neurofibromas. Pediatr Blood Cancer. 2013 Mar;60(3):396-401. doi: 10.1002/pbc.24281. Epub 2012 Sep 7. PMID 22961690
- [Background] Lasater EA, Bessler WK, Mead LE, Horn WE, Clapp DW, Conway SJ, Ingram DA, Li F. Nf1+/- mice have increased neointima formation via hyperactivation of a Gleevec sensitive molecular pathway. Hum Mol Genet. 2008 Aug 1;17(15):2336-44. doi: 10.1093/hmg/ddn134. Epub 2008 Apr 28. PMID 18442999
- [Background] McCormick F. Ras signaling and NF1. Curr Opin Genet Dev. 1995 Feb;5(1):51-5. doi: 10.1016/s0959-437x(95)90053-5. PMID 7749326
- [Background] Sherman LS, Atit R, Rosenbaum T, Cox AD, Ratner N. Single cell Ras-GTP analysis reveals altered Ras activity in a subpopulation of neurofibroma Schwann cells but not fibroblasts. J Biol Chem. 2000 Sep 29;275(39):30740-5. doi: 10.1074/jbc.M001702200. PMID 10900196
- [Background] Downward J. Targeting RAS signalling pathways in cancer therapy. Nat Rev Cancer. 2003 Jan;3(1):11-22. doi: 10.1038/nrc969. PMID 12509763
- [Background] Weiss B, Bollag G, Shannon K. Hyperactive Ras as a therapeutic target in neurofibromatosis type 1. Am J Med Genet. 1999 Mar 26;89(1):14-22. PMID 10469432
- [Background] Wu J, Dombi E, Jousma E, Scott Dunn R, Lindquist D, Schnell BM, Kim MO, Kim A, Widemann BC, Cripe TP, Ratner N. Preclincial testing of sorafenib and RAD001 in the Nf(flox/flox) ;DhhCre mouse model of plexiform neurofibroma using magnetic resonance imaging. Pediatr Blood Cancer. 2012 Feb;58(2):173-80. doi: 10.1002/pbc.23015. Epub 2011 Feb 11. PMID 21319287
- [Background] Kissil JL, Blakeley JO, Ferner RE, Huson SM, Kalamarides M, Mautner VF, McCormick F, Morrison H, Packer R, Ramesh V, Ratner N, Rauen KA, Stevenson DA, Hunter-Schaedle K, North K. What's new in neurofibromatosis? Proceedings from the 2009 NF Conference: new frontiers. Am J Med Genet A. 2010 Feb;152A(2):269-83. doi: 10.1002/ajmg.a.33189. PMID 20082461
- [Background] Yang FC, Ingram DA, Chen S, Zhu Y, Yuan J, Li X, Yang X, Knowles S, Horn W, Li Y, Zhang S, Yang Y, Vakili ST, Yu M, Burns D, Robertson K, Hutchins G, Parada LF, Clapp DW. Nf1-dependent tumors require a microenvironment containing Nf1+/-- and c-kit-dependent bone marrow. Cell. 2008 Oct 31;135(3):437-48. doi: 10.1016/j.cell.2008.08.041. PMID 18984156
- [Background] Jessen WJ, Miller SJ, Jousma E, Wu J, Rizvi TA, Brundage ME, Eaves D, Widemann B, Kim MO, Dombi E, Sabo J, Hardiman Dudley A, Niwa-Kawakita M, Page GP, Giovannini M, Aronow BJ, Cripe TP, Ratner N. MEK inhibition exhibits efficacy in human and mouse neurofibromatosis tumors. J Clin Invest. 2013 Jan;123(1):340-7. doi: 10.1172/JCI60578. Epub 2012 Dec 10. PMID 23221341
- [Background] Chang T, Krisman K, Theobald EH, Xu J, Akutagawa J, Lauchle JO, Kogan S, Braun BS, Shannon K. Sustained MEK inhibition abrogates myeloproliferative disease in Nf1 mutant mice. J Clin Invest. 2013 Jan;123(1):335-9. doi: 10.1172/JCI63193. Epub 2012 Dec 10. PMID 23221337
- [Background] Nutakki K, Hingtgen CM, Monahan P, Varni JW, Swigonski NL. Development of the adult PedsQL neurofibromatosis type 1 module: initial feasibility, reliability and validity. Health Qual Life Outcomes. 2013 Feb 21;11:21. doi: 10.1186/1477-7525-11-21. PMID 23432799
- [Background] Rosser T, Packer RJ. Neurofibromas in children with neurofibromatosis 1. J Child Neurol. 2002 Aug;17(8):585-91; discussion 602-4, 646-51. doi: 10.1177/088307380201700808. PMID 12403557
- [Background] Le LQ, Parada LF. Tumor microenvironment and neurofibromatosis type I: connecting the GAPs. Oncogene. 2007 Jul 12;26(32):4609-16. doi: 10.1038/sj.onc.1210261. Epub 2007 Feb 12. PMID 17297459
- [Background] Prada CE, Jousma E, Rizvi TA, Wu J, Dunn RS, Mayes DA, Cancelas JA, Dombi E, Kim MO, West BL, Bollag G, Ratner N. Neurofibroma-associated macrophages play roles in tumor growth and response to pharmacological inhibition. Acta Neuropathol. 2013 Jan;125(1):159-68. doi: 10.1007/s00401-012-1056-7. Epub 2012 Oct 26. PMID 23099891
- [Background] Wolkenstein P, Zeller J, Revuz J, Ecosse E, Leplege A. Quality-of-life impairment in neurofibromatosis type 1: a cross-sectional study of 128 cases. Arch Dermatol. 2001 Nov;137(11):1421-5. doi: 10.1001/archderm.137.11.1421. PMID 11708944
- See also: A phase 1 study of mitogen activated protein kinase (MEK) 1 inhibitor AZD6244 hydrogen sulfate (selumetinib sulfate) in children with neurofibromatosis type 1 (NF1) and inoperable plexiform neurofibromas (PN) — http://clinicaltrials.gov/show/NCT01362803
- See also: Chow, L., et al. "A first in human dose-ranging study to assess the pharmacokinetics, pharmacodynamics, and toxicities of the MEK inhibitor, ARRY-142886 (AZD6244), in patients with advanced solid malignancies." CLINICAL CANCER RESEARCH. Vol. 11. No.24 — https://scholar.google.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Open Label Study of Binimetinib (MEK162): Subjects (≥ 18 years) (Stratum A) will receive a course of binimetinib by mouth twice a day (12 hours apart) of 45 mg/dose. Duration of each course is 4 weeks. After 8 courses, subjects will receive additional courses if MRI results showed at least 15% reduction in volume of the target tumor. Subjects can continue on therapy and will be evaluated at the end of 12 courses. Subjects who have ≥ 20% reduction in volume of the target tumor according to the MRI results can continue therapy up to an additional year (maximum of 24 total courses). Subjects who have not met the tumor reduction at the specified times will be removed from the study therapy. Subjects will be carefully monitored for toxicities associated with binimetinib.
  Recruitment of subjects 1 - 17 years of age (Stratum B) is currently available. The pediatric maximum tolerated dose (MTD) of binimetinib the pediatric patients (Statum B) was established by a phase 1 study (NCT022).
  Binimetinib: Adult subjects (18 years and older) will receive binimetinib by mouth twice daily of 45mg/dose. Pediatric subjects (1-17 years of age) are being treated on the pediatric MTD established by a phase I study (NCT02285439).
Period: Overall Study
Arm/Group | Open Label Study of Binimetinib (MEK162)
Started | 45
Completed | 19
Not Completed | 26
Not completed — <15% reduction in target tumor volume from baseline after Course 8 of therapy | 3
Not completed — <20% reduction in target tumor volume from baseline after Course 12 of therapy | 4
Not completed — Treatment delay > 21 days | 2
Not completed — Refusal of further protocol therapy by subject/parent/guardian | 6
Not completed — Non-compliance that in the opinion of the investigator does not allow for ongoing participation | 5
Not completed — Binimetinib-related toxicity requiring removal from protocol therapy | 3
Not completed — Subject Relocation Due to Covid Restrictions | 1
Not completed — More than 1 Reason | 2

BASELINE CHARACTERISTICS:
Population: Binimetinib: Adult subjects (18 years and older) will receive binimetinib by mouth twice daily of 45mg/dose. Pediatric subjects (1-17 years of age) are being treated on the pediatric MTD established by a phase I study (NCT02285439).
Arm/Group | Open Label Study of Binimetinib (MEK162)
Number analyzed (Participants) | 45
Age, Continuous [Median (Full Range); unit: Years] | 19 [2 to 55]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 39
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 28
  More than one race | 2
  Unknown or Not Reported | 10
Region of Enrollment [Number; unit: participants]
  United States | 45
Number of Participants [Count of Participants; unit: Participants] | 45

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline Target Tumor Volume at 12 Months
Description: To determine the objective response defined as 20% or greater tumor volume reduction. Patients will undergo volumetric assays of their target PN using MRI.
Time Frame: Approximately 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Open Label Study of Binimetinib (MEK162)
Number analyzed (Participants) | 44
Participants
  Met Objective Response | 27
  Did Not Meet Objective Response | 17

2. Secondary Outcome: Incidence of Treatment-Emergent Adverse Events
Description: To evaluate the toxicity of protracted binimetinib administration in this patient population. Subjects will be monitored continuously for adverse events and serious adverse events throughout the study.
Time Frame: Up to 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Open Label Study of Binimetinib (MEK162)
Number analyzed (Participants) | 45
Participants | 45

ADVERSE EVENTS:
Time Frame: 24 Months
Arm/Group | Open Label Study of Binimetinib (MEK162)
All-Cause Mortality (participants affected / at risk) | 0/45
Serious Adverse Events (participants affected / at risk) | 11/45
Other Adverse Events (participants affected / at risk) | 45/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open Label Study of Binimetinib (MEK162) (N=45)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (5)
Diarrhea (Gastrointestinal disorders) | 1 (2)
Gastric Hemorrhage (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Anaphylaxis (Immune system disorders) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1)
Skin Infection (Infections and infestations) | 1 (1)
Weight Loss (Metabolism and nutrition disorders) | 1 (1)
Suicide attempt (Psychiatric disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open Label Study of Binimetinib (MEK162) (N=45)
Anemia (Blood and lymphatic system disorders) | 16 (36)
Cardiac disorders - Other, Non-Specific St And T-Wave Abnormalities (Cardiac disorders) | 1 (1)
Cardiac disorders - Other, Nonspecific T Wave Abnormality (Cardiac disorders) | 1 (1)
Cardiac disorders - Other, Specify, Electrocardiogram T Wave Abnormal (Cardiac disorders) | 2 (2)
Cardiac disorders - Other, Systolic Murmur (Cardiac disorders) | 1 (1)
Cardiac disorders - Other, Tachycardia (Cardiac disorders) | 1 (1)
Conduction disorder (Cardiac disorders) | 1 (1)
Pulmonary Valve Disease (Cardiac disorders) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 4 (8)
Ventricular Arrhythmia (Cardiac disorders) | 1 (1)
Ear and labyrinth disorders - Other, Mastoid Effusion (Ear and labyrinth disorders) | 1 (1)
External Ear Inflammation (Ear and labyrinth disorders) | 1 (1)
Endocrine disorders - Other, Increased Intolerance To Heat And Humidity (Endocrine disorders) | 1 (1)
Blurred Vision (Eye disorders) | 2 (3)
Conjunctivitis (Eye disorders) | 2 (2)
Corneal ulcer (Ear and labyrinth disorders) | 1 (1)
Dry Eye (Eye disorders) | 1 (1)
Eye disorders - Other, Blepharitis (Eye disorders) | 1 (1)
Eye disorders - Other, Central Lenticular Opacities (Eye disorders) | 1 (1)
Eye disorders - Other, Erythema (Eye disorders) | 1 (1)
Eye disorders - Other, Macular Edema (Eye disorders) | 1 (1)
Eye disorders - Other, Optic Disk Swelling With Peripapillary Hemorrhages (Eye disorders) | 1 (1)
Eye pain (Eye disorders) | 1 (2)
Floaters (Eye disorders) | 1 (1)
Keratitis (Eye disorders) | 2 (3)
Scleral disorder (Eye disorders) | 1 (1)
Abdominal Distention (Gastrointestinal disorders) | 1 (2)
Abdominal Pain (Gastrointestinal disorders) | 13 (28)
Cheilitis (Gastrointestinal disorders) | 2 (3)
Constipation (Gastrointestinal disorders) | 10 (11)
Diarrhea (Gastrointestinal disorders) | 28 (77)
Dry Mouth (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 5 (8)
Emesis (Gastrointestinal disorders) | 1 (1)
Fecal Incontinence (Gastrointestinal disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 4 (4)
Gastric Hemorrhage (Gastrointestinal disorders) | 1 (1)
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 2 (3)
Gastrointestinal disorders - Other, Specify Tooth Loss (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorders - Other, Tooth Pain (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorders - Other, Cecal Volvulus (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorders Gastrointestinal disorders - Other, Gastroenteritis (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorders - Other, Mouth Sore (Gastrointestinal disorders) | 2 (2)
Gastrointestinal pain (Gastrointestinal disorders) | 1 (1)
Hemorrhoidal Hemorrhage (Gastrointestinal disorders) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 7 (15)
Nausea (Gastrointestinal disorders) | 27 (52)
Small Intestinal Obstruction (Gastrointestinal disorders) | 1 (1)
Stomach Pain (Gastrointestinal disorders) | 4 (5)
Vomiting (Gastrointestinal disorders) | 23 (66)
Chills (General disorders) | 5 (5)
Edema Face (General disorders) | 7 (12)
Edema Limbs (General disorders) | 11 (26)
Edema Trunk (Gastrointestinal disorders) | 1 (2)
Facial Pain (General disorders) | 1 (1)
Fatigue (General disorders) | 21 (36)
Fever (General disorders) | 11 (21)
Flu Like Symptoms (General disorders) | 3 (3)
General Disorders and Administration Site Conditions - Other, Bleeding Gums (General disorders) | 1 (1)
Irritability (General disorders) | 2 (3)
Localized Edema (General disorders) | 3 (10)
Malaise (General disorders) | 2 (2)
Non-Cardiac Chest Pain (General disorders) | 4 (5)
Pain (General disorders) | 3 (3)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Allergic Reaction (Immune system disorders) | 2 (3)
Eye Infection (Infections and infestations) | 1 (1)
Infections And Infestations, Other, Folliculitis (Infections and infestations) | 1 (2)
Infections and infestations - Other, BK Virus (Infections and infestations) | 1 (1)
Infections and infestations - Other, Covid-19 (Infections and infestations) | 2 (2)
Infections and infestations - Other, Gastroenteritis (Infections and infestations) | 1 (1)
Nail Infection (Infections and infestations) | 1 (1)
Otitis Externa (Infections and infestations) | 3 (3)
Otitis Media (Infections and infestations) | 3 (3)
Papulopustular rash (Infections and infestations) | 4 (4)
Paronychia (Infections and infestations) | 18 (52)
Pharyngitis (Infections and infestations) | 2 (2)
Rash pustular (Infections and infestations) | 1 (2)
Sinusitis (Infections and infestations) | 1 (1)
Skin Infection (Infections and infestations) | 13 (21)
Upper Respiratory Infection (Infections and infestations) | 4 (4)
Urinary Tract Infection (Infections and infestations) | 2 (3)
Vaginal Infection (Infections and infestations) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 1 (1)
Burn (Injury, poisoning and procedural complications) | 1 (2)
Wound Complication (Injury, poisoning and procedural complications) | 1 (1)
Alanine Aminotransferase Increased (Investigations) | 12 (32)
Alkaline Phosphatase Increased (Investigations) | 4 (6)
Aspartate Aminotransferase Increased (Investigations) | 23 (43)
Blood bilirubin increased (Investigations) | 4 (8)
CPK increased (Investigations) | 33 (96)
Creatinine Increased (Investigations) | 2 (5)
Ejection fraction decreased (Investigations) | 3 (4)
Electrocardiogram Qt Corrected Interval Prolonged (Investigations) | 1 (1)
Growth Hormone Abnormal (Investigations) | 1 (1)
Hemoglobin Increased (Investigations) | 1 (2)
Investigations - Other, Absolute Lymphocyte Count Increased (Investigations) | 1 (1)
Investigations - Other, Absolute Neutrophil Count Decreased (Investigations) | 3 (5)
Investigations - Other, Creatine Kinase Increased (Investigations) | 1 (2)
Investigations - Other, Lactate Dehydrogenase Increased (Investigations) | 1 (1)
Investigations - Other, Partial Thromboplastin Time Prolonged (Investigations) | 1 (2)
Lipase Increased (Investigations) | 1 (1)
Lymphocyte Count Decreased (Investigations) | 4 (6)
Neutrophil Count Decreased (Investigations) | 7 (13)
Platelet Count Decreased (Investigations) | 5 (9)
Weight Gain (Investigations) | 8 (22)
Weight Loss (Investigations) | 3 (7)
White Blood Cell Decreased (Investigations) | 7 (11)
Anorexia (Metabolism and nutrition disorders) | 6 (7)
Dehydration (Metabolism and nutrition disorders) | 6 (7)
Hypercalcemia (Metabolism and nutrition disorders) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (6)
Hyperkalemia (Metabolism and nutrition disorders) | 5 (10)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 3 (3)
Hypoalbuminemia (Metabolism and nutrition disorders) | 12 (23)
Hypocalcemia (Metabolism and nutrition disorders) | 7 (13)
Hypoglycemia (Metabolism and nutrition disorders) | 4 (12)
Hypokalemia (Metabolism and nutrition disorders) | 7 (16)
Hypomagnesemia (Metabolism and nutrition disorders) | 3 (4)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 4 (5)
Metabolism And Nutrition Disorders - Other, Decreased Appetite (Metabolism and nutrition disorders) | 1 (1)
Metabolism And Nutrition Disorders - Other, Hyperphosphatemia (Metabolism and nutrition disorders) | 3 (5)
Metabolism And Nutrition Disorders - Other, Total Protein Decreased (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Back Pain (Musculoskeletal and connective tissue disorders) | 4 (5)
Bone Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Generalized Muscle Weakness (Musculoskeletal and connective tissue disorders) | 5 (9)
Lordosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle weakness trunk (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal And Connective Tissue Disorder - Other, Pain Head/Neck/Extremities (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal And Connective Tissue Disorders - Other, Leg Cramps (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal and connective tissue disorders - Other, Joint Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 7 (9)
Neck Pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 5 (6)
Cognitive Disturbance (Nervous system disorders) | 2 (2)
Dizziness (Nervous system disorders) | 9 (12)
Dysgeusia (Nervous system disorders) | 2 (2)
Headache (Nervous system disorders) | 11 (18)
Memory Impairment (Nervous system disorders) | 1 (1)
Paresthesia (Nervous system disorders) | 3 (3)
Presyncope (Nervous system disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 2 (2)
Agitation (Psychiatric disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 3 (3)
Depression (Psychiatric disorders) | 4 (5)
Insomnia (Psychiatric disorders) | 6 (6)
Cystitis Noninfective (Renal and urinary disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 4 (4)
Proteinuria (Renal and urinary disorders) | 2 (3)
Renal And Urinary Disorders - Other, Dysuria (Renal and urinary disorders) | 1 (1)
Renal And Urinary Disorders - Other, Elevated Bun (Renal and urinary disorders) | 1 (1)
Renal And Urinary Disorders - Other, Weak Urine Stream (Renal and urinary disorders) | 1 (1)
Urinary Incontinence (Renal and urinary disorders) | 1 (1)
Urinary Retention (Renal and urinary disorders) | 1 (1)
Urinary Urgency (Renal and urinary disorders) | 2 (5)
Menorrhagia (Reproductive system and breast disorders) | 1 (2)
Reproductive System And Breast Disorders - Other, Breast Lump (Reproductive system and breast disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (8)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6 (8)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Laryngeal Inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Laryngeal Obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 2 (4)
Postnasal Drip (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Respiratory, Thoracic And Mediastinal Disorders - Other, Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 4 (6)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 15 (19)
Dry Skin (Skin and subcutaneous tissue disorders) | 19 (28)
Erythema Multiforme (Skin and subcutaneous tissue disorders) | 1 (1)
Palmar-Plantar Erythrodysesthesia Syndrome (Skin and subcutaneous tissue disorders) | 1 (1)
Periorbital Edema (Skin and subcutaneous tissue disorders) | 3 (3)
Photosensitivity (Skin and subcutaneous tissue disorders) | 3 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 9 (12)
Purpura (Skin and subcutaneous tissue disorders) | 1 (3)
Rash acneiform (Skin and subcutaneous tissue disorders) | 38 (53)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 14 (22)
Scalp Pain (Skin and subcutaneous tissue disorders) | 2 (3)
Skin Atrophy (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other, Achromotrichia (Skin and subcutaneous tissue disorders) | 2 (2)
Skin and subcutaneous tissue disorders - Other, Diaper Dermatitis (Skin and subcutaneous tissue disorders) | 1 (5)
Skin and subcutaneous tissue disorders - Other, Eczema (Skin and subcutaneous tissue disorders) | 2 (2)
Skin and subcutaneous tissue disorders - Other, Erythemous Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other, Hair Color Changes (Skin and subcutaneous tissue disorders) | 4 (4)
Skin and subcutaneous tissue disorders - Other, Insect Bites (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other, Mottled Skin (Skin and subcutaneous tissue disorders) | 2 (2)
Skin and subcutaneous tissue disorders - Other, Papulopustular Rash (Skin and subcutaneous tissue disorders) | 2 (3)
Skin and subcutaneous tissue disorders - Other, Petechiae (Skin and subcutaneous tissue disorders) | 1 (2)
Skin and subcutaneous tissue disorders - Other, Seborrheic Dermatitis (Skin and subcutaneous tissue disorders) | 5 (12)
Skin and subcutaneous tissue disorders - Other, Sore on Foot (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other, Sunburn (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other, Unspecified Rash (Skin and subcutaneous tissue disorders) | 2 (3)
Hypertension (Vascular disorders) | 7 (10)
Hypotension (Vascular disorders) | 1 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-02-16): https://cdn.clinicaltrials.gov/large-docs/06/NCT03231306/Prot_SAP_000.pdf
  • Informed Consent Form (2023-02-17): https://cdn.clinicaltrials.gov/large-docs/06/NCT03231306/ICF_001.pdf